CLINICAL TRIAL: NCT05646927
Title: Effect of Child Preference for Parental Selection During Induction in Children Undergoing Elective Day Case Surgery
Brief Title: Effect of Child Preference for Parental Selection During Induction
Status: Completed | Type: Observational
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 09-2022/04
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2022-12

CONDITIONS: Anxiety State; Child Behavior
Keywords: day- case surgery; anxiety; children
MeSH Terms: conditions — Anxiety Disorders; Child Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Child Preference: The children will prefer parents (mother or father) who will accompany them in the preoperative holding area and at induction.
  Interventions: Procedure: Selection of parent(mother or father) according to children preference
- Group None: The parent of the children who will accompany them during the perioperative period will be determined according to randomization.
  Interventions: Procedure: Selection of parent(mother or father) according to randomization

INTERVENTIONS:
Procedure: Selection of parent(mother or father) according to children preference — The parent who will accompany the child during the perioperative period will be determined by children preference
  Groups: Group Child Preference
Procedure: Selection of parent(mother or father) according to randomization — The parent who will accompany the child during the perioperative period will be determined by randomization.
  Groups: Group None

SUMMARY:
Induction of anesthesia can be distressing both for children and their parents. Nonpharmacological behavioral interventions can reduce the anxiety of children without significant adverse effects as seen with sedative drugs. has not been documented.

The aim of this study will be to evaluate the effect of children's preference on parental selection during the induction of anesthesia on children and parental anxiety during the perioperative period.

DETAILED DESCRIPTION:
Anesthetic induction can be one of the most stressful experiences for the child during the perioperative period, with almost 50% of the children showing significant anxiety. . To minimize the effect of anxiety, several methods have been adopted, such as the introduction of day-case surgery, parental presence at the induction of anesthesia, distractions and the use of pharmacological agents like midazolam to reduce anxiety.

Although the effect of parental presence on the anxiety of children and parents was studied in various studies. Whether the children's choice of parental selection affects anxiety is not studied yet. In this study, we will evaluate the anxiety of children by using mYPAS .

ELIGIBILITY:
Inclusion Criteria:

* 80 children of both sex, aged 4-15 years with ASA physical Status I-II will be enrolled

Exclusion Criteria:

1. Mentally challenged
2. Deaf Child
3. Cerebral Palsy
4. Premedicated Child
5. Language Problem
6. Unco-operative
7. Previous surgery or anesthesia history

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 80 children of both sex, aged 4-8 years with ASA physical Status I-II will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Modified Yale Preoperative Anxiety Scale (mYPAS) of the children undergoing elective surgery under general anesthesia. | Perioperative period
  The mYPAS will be used to evaluate the anxiety level of children. The mYPAS is an observational measure of preoperative anxiety consisting of 27 items in 5 domains (activity, emotional expressivity, state of arousal, vocalization, and use of parents). The adjusted mYPAS total score ranges from 22.9 to 100, with higher scores indicating greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Yucedag, Assist Prof, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)

REFERENCES:
- [Derived] Fatih Y, Arife S, Aysegul B, Betul B. The Effect of Child Preference for Parental Selection on Pediatric Anxiety During Induction in Children Undergoing Elective Day Case Surgery. J Perianesth Nurs. 2024 Jun;39(3):397-402. doi: 10.1016/j.jopan.2023.08.021. Epub 2023 Dec 5. PMID 38054915